CLINICAL TRIAL: NCT04497350
Title: A Blinded, Randomized Trial Comparing the Effects of Transcranial Magnetic Stimulation and Theta Burst Stimulation in Patients With Major Depressive Disorder
Brief Title: Transcranial Magnetic Stimulation vs Theta Burst Stimulation in Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20193262
Record Dates: First submitted 2020-06-16; First posted 2020-08-04 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder
Keywords: transcranial magnetic stimulation; theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a single-site, randomized, blinded, clinical trial comparing the efficacy of transcranial magnetic stimulation (TMS) and intermittent theta burst stimulation (iTBS) in subjects with treatment refractory depression (trMDD). The study will recruit 30 subjects, all suffering from treatment refractory depression (trMDD). Half of the subjects (15) will be randomized to the TMS treatment group, while the other half will be assigned to the iTBS treatment group. The randomization ratio will be 1:1.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Magnetic Stimulation (Experimental): All patients are required to have an advanced MRI of the brain including a structural T1, volume measurements of various brain regions, ASL, and BOLD sequences. Patients will also undergo an in-scanner task designed to activate key neurofunctional regions of interest.
  Interventions: Device: Transcranial Magnetic Stimulation
- Theta Burst Stimulation (Experimental): All patients are required to have an advanced MRI of the brain including a structural T1, volume measurements of various brain regions, ASL, and BOLD sequences. Patients will also undergo an in-scanner task designed to activate key neurofunctional regions of interest.
  Interventions: Device: Theta Burst Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — 5,000 pulses (120-140% MT, continuous temperature of 24C) will be delivered per session (see Appendix A for timing parameters). Patients will have one TMS session per day, five days a week, until their treatment is completed (approximately four weeks).
  Arms: Transcranial Magnetic Stimulation
Device: Theta Burst Stimulation — One session of iTBS will deliver 1,800 pulses (120-140% MT, continuous temperature of 22ºC) over an 9-minute-40-second period. The minimum break period between iTBS sessions is 25 minutes.
  Arms: Theta Burst Stimulation

SUMMARY:
The purpose of this study is to investigate the differences in efficacy between transcranial magnetic stimulation (TMS) and intermittent theta burst stimulation (iTBS) treatment in subjects suffering from major depressive disorder.

DETAILED DESCRIPTION:
Up to 30 patients of any gender aged from 18 to 70 years old will be recruited for inclusion once candidacy has been established by screening criteria.

Once recruited, patients will be randomly assigned to the TMS treatment group or the iTBS treatment group. Patients will be blinded to their group assignment, but will be informed of their assignment upon the final outcome measure collection timepoint (e.g., 1 month post-treatment). Patients who failed to respond by 1-month post iTBS or TMS treatment will be allowed to cross-over into the other treatment group and will be re-enrolled into the study.

For patients assigned to the TMS treatment group, the treatment protocol will consist of 20 sessions of TMS treatment. Each TMS session will deliver 5,000 pulses (120-140% MT, continuous temperature of 24C) over an 61 minute, 51 second time period. Patients will have one TMS session per day, five days a week, until their treatment is completed (approximately four weeks). Upon completion, the patient's depressive symptomatology and severity will be assessed using the same outcome measures used at baseline.

For patients assigned to the iTBS treatment group, the treatment protocol will consist of 20 sessions of iTBS treatment. Each iTBS session will deliver 1,800 pulses (120-140% MT, continuous temperature of 24C) over an 9-minute-40-second period. Patients will have up to four iTBS sessions per day, five days a week, until their treatment is completed (approximately 1 week). Upon completion, the patient's depressive symptomatology and severity will be assessed using the same outcome measures used at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder
* Score greater than 13 on the Beck Depression Inventory
* Failure to remit with 3 antidepressants
* At least 18 years of age
* Must be willing to comply with the study protocol
* English Proficiency

Exclusion Criteria:

* Hepatic impairment
* Significant cytopenia
* Cardiovascular, cerebrovascular, and peripheral vascular arterial thrombosis
* Advanced terminal illness
* Any active cancer or chemotherapy
* Bone marrow disease
* Neurodegenerative diseases
* Myeloproliferative disorders
* Sickle cell disease
* Subjects with scalp rash or open wounds on the scalp
* Women who are pregnant, may become pregnant, or are breastfeeding
* Subjects unable to give informed consent or in vulnerable categories, such as prisoners
* Subjects who would not be able to lay down without excessive movement
* Recent surgery or dental work within 3 months of the scheduled procedure
* Not English Proficient
* Advanced stages of any terminal illness or any active cancer that requires chemotherapy
* History of epilepsy or seizure, or history of such in first degree relative
* An increased risk of seizure for any reason
* Stents in the neck or brain
* Aneurysm clips or coils
* Metal devices/objects in or near the head
* Metallic implants near the ears and eyes
* Facial tattoos with metallic or magnetic-sensitive ink
* Comorbid psychiatric conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-II) | 1 month
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Patient Depression Questionnaire (PDQ-9) | 1 month
  The PDQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.
Hamilton Depression Rating Scale (HAM-D) | 1 month
  The HAM-D is a 17-item, interview style questionnaire. A trained staff member administers this form to a patient and scores the patients' responses on a scale of "0" (symptom absent) to "4" (most severe option per symptom). A higher total score indicates a more severe level of depression. The maximum possible score is 50 points. A change in score of at least 30% is considered clinically meaningful.
Global Rating of Change (GRC) | 1 month
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II) | 2 months
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Patient Depression Questionnaire (PDQ-9) | 2 months
  The PDQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.
Hamilton Depression Rating Scale (HAM-D) | 2 months
  The HAM-D is a 17-item, interview style questionnaire. A trained staff member administers this form to a patient and scores the patients' responses on a scale of "0" (symptom absent) to "4" (most severe option per symptom). A higher total score indicates a more severe level of depression. The maximum possible score is 50 points. A change in score of at least 30% is considered clinically meaningful.
Global Rating of Change (GRC) | 2 months
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon E Jordan, M.D., Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be made publicly available due to ethical and privacy concerns. Anonymized data will be available upon reasonable request from any qualified investigator.

REFERENCES:
- [Background] Ferrari AJ, Charlson FJ, Norman RE, Patten SB, Freedman G, Murray CJ, Vos T, Whiteford HA. Burden of depressive disorders by country, sex, age, and year: findings from the global burden of disease study 2010. PLoS Med. 2013 Nov;10(11):e1001547. doi: 10.1371/journal.pmed.1001547. Epub 2013 Nov 5. PMID 24223526
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Setiawan E, Attwells S, Wilson AA, Mizrahi R, Rusjan PM, Miler L, Xu C, Sharma S, Kish S, Houle S, Meyer JH. Association of translocator protein total distribution volume with duration of untreated major depressive disorder: a cross-sectional study. Lancet Psychiatry. 2018 Apr;5(4):339-347. doi: 10.1016/S2215-0366(18)30048-8. Epub 2018 Feb 26. PMID 29496589
- [Background] Drevets WC, Savitz J, Trimble M. The subgenual anterior cingulate cortex in mood disorders. CNS Spectr. 2008 Aug;13(8):663-81. doi: 10.1017/s1092852900013754. PMID 18704022
- [Background] Lozano AM, Mayberg HS, Giacobbe P, Hamani C, Craddock RC, Kennedy SH. Subcallosal cingulate gyrus deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2008 Sep 15;64(6):461-7. doi: 10.1016/j.biopsych.2008.05.034. Epub 2008 Jul 18. PMID 18639234
- [Background] Mayberg HS, Liotti M, Brannan SK, McGinnis S, Mahurin RK, Jerabek PA, Silva JA, Tekell JL, Martin CC, Lancaster JL, Fox PT. Reciprocal limbic-cortical function and negative mood: converging PET findings in depression and normal sadness. Am J Psychiatry. 1999 May;156(5):675-82. doi: 10.1176/ajp.156.5.675. PMID 10327898
- [Background] Botteron KN, Raichle ME, Drevets WC, Heath AC, Todd RD. Volumetric reduction in left subgenual prefrontal cortex in early onset depression. Biol Psychiatry. 2002 Feb 15;51(4):342-4. doi: 10.1016/s0006-3223(01)01280-x. PMID 11958786
- [Background] Yucel K, McKinnon M, Chahal R, Taylor V, Macdonald K, Joffe R, Macqueen G. Increased subgenual prefrontal cortex size in remitted patients with major depressive disorder. Psychiatry Res. 2009 Jul 15;173(1):71-6. doi: 10.1016/j.pscychresns.2008.07.013. Epub 2009 May 21. PMID 19464154
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Daskalakis ZJ, Christensen BK, Fitzgerald PB, Chen R. Transcranial magnetic stimulation: a new investigational and treatment tool in psychiatry. J Neuropsychiatry Clin Neurosci. 2002 Fall;14(4):406-15. doi: 10.1176/jnp.14.4.406. PMID 12426408
- [Background] Eldaief MC, Press DZ, Pascual-Leone A. Transcranial magnetic stimulation in neurology: A review of established and prospective applications. Neurol Clin Pract. 2013 Dec;3(6):519-526. doi: 10.1212/01.CPJ.0000436213.11132.8e. PMID 24353923
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Eldaief MC, Halko MA, Buckner RL, Pascual-Leone A. Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner. Proc Natl Acad Sci U S A. 2011 Dec 27;108(52):21229-34. doi: 10.1073/pnas.1113103109. Epub 2011 Dec 12. PMID 22160708
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Background] Strafella AP, Paus T, Barrett J, Dagher A. Repetitive transcranial magnetic stimulation of the human prefrontal cortex induces dopamine release in the caudate nucleus. J Neurosci. 2001 Aug 1;21(15):RC157. doi: 10.1523/JNEUROSCI.21-15-j0003.2001. PMID 11459878
- [Background] Cho SS, Strafella AP. rTMS of the left dorsolateral prefrontal cortex modulates dopamine release in the ipsilateral anterior cingulate cortex and orbitofrontal cortex. PLoS One. 2009 Aug 21;4(8):e6725. doi: 10.1371/journal.pone.0006725. PMID 19696930
- [Background] Di Lazzaro V, Pilato F, Dileone M, Profice P, Oliviero A, Mazzone P, Insola A, Ranieri F, Meglio M, Tonali PA, Rothwell JC. The physiological basis of the effects of intermittent theta burst stimulation of the human motor cortex. J Physiol. 2008 Aug 15;586(16):3871-9. doi: 10.1113/jphysiol.2008.152736. Epub 2008 Jun 19. PMID 18566003
- [Background] Larson J, Wong D, Lynch G. Patterned stimulation at the theta frequency is optimal for the induction of hippocampal long-term potentiation. Brain Res. 1986 Mar 19;368(2):347-50. doi: 10.1016/0006-8993(86)90579-2. PMID 3697730
- [Background] Suppa A, Huang YZ, Funke K, Ridding MC, Cheeran B, Di Lazzaro V, Ziemann U, Rothwell JC. Ten Years of Theta Burst Stimulation in Humans: Established Knowledge, Unknowns and Prospects. Brain Stimul. 2016 May-Jun;9(3):323-335. doi: 10.1016/j.brs.2016.01.006. Epub 2016 Jan 27. PMID 26947241
- [Background] Kearney-Ramos TE, Dowdle LT, Lench DH, Mithoefer OJ, Devries WH, George MS, Anton RF, Hanlon CA. Transdiagnostic Effects of Ventromedial Prefrontal Cortex Transcranial Magnetic Stimulation on Cue Reactivity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jul;3(7):599-609. doi: 10.1016/j.bpsc.2018.03.016. Epub 2018 Apr 10. PMID 29776789
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011